CLINICAL TRIAL: NCT06003374
Title: Extended Hip Ultrasound as Anew Protocol for Septic Hip in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dalia Khaled Mostafa Mohamed, Resident doctor at diagnostic radiology department at assuit univerity, Assiut University
Other Study IDs: US in pediateric septic hip.
Record Dates: First submitted 2022-12-17; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-06

CONDITIONS: Septic Arthritis
MeSH Terms: conditions — Arthritis, Infectious | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound — At international protocol U/S examination is performed from an anterior approach, with the transducer in a sagittal plane parallel to the femoral neck. The patients are positioned supine with the hips in neutral position. Also a coronal view is performed from the lateral approach. Establish a new protocol in the MSK unit to perform hip US,
  * adductor view: flexion, abduction and lateral rotation of the hip joint with viewing the hip via adductor muscle group.
  * gluteal view: posterior approach of the hip joint via gluteal region with the patient lying on the contralateral examined hip.
  Psoas and thigh views: US examination of psoas and quadriceps muscles to exclude the presence of absecess .
  -finally US guided aspiration under complete a septic condition.

SUMMARY:
To establish a new protocol in order to increase ultrasound diagnostic accuracy of pediatrics presented with signs of septic hip .

DETAILED DESCRIPTION:
Septic arthritis is a severe life and function threatening condition with a 1-year mortality rate of up to 10% and residual functional impairments in 30% to 50% of cases . Pediatric Septic Hip Arthritis is an intra-articular infection in children that peaks in the first few years of life. The incidence of septic arthritis is low, with about 4-5 per 100000 child annually with about 50% of cases occur in children younger than 2 years of age with gender affection in male > female (2:1 ratio). The hip joint involved in about 35% of all cases of septic arthritis. Imaging studies contribute crucially to the optimal management of septic arthritis, thereby diminishing the risk of permanent functional loss .At present; magnetic resonance imaging (MRI) is the most informative method. Thus, MRI assesses the severity of the synovitis and can detect a joint effusion, bone and/or cartilage destruction, an abscess, and/or bone edema. MRI had 75% specificity and nearly 100% sensitivity for diagnosing concomitant abscess formation, cellulitis, or myositis . Disadvantages of MRI are high cost and limited availability on an emergency basis in some settings , Ultrasonography of the bone and joints has been developing at a fast pace in recent years. Ultrasonography is currently used in the management of septic arthritis to confirm the presence of a joint effusion and to guide the joint aspiration or synovial biopsy, particularly when the effusion is small or the joint deep (e.g., hip). Ultrasonography has high sensitivity and specificity for joint effusions .The difficulty of applying hip MRI in pediatric age group patients especially neonates make challenge in the proper management of acute septic hip arthritis .the study aim to apply a new protocol in diagnosis of septic hip in children by doing extended hip ultrasound included psoas and quadriceps muscles.

ELIGIBILITY:
Inclusion Criteria:

* Neonates, infants and children presented with suspected septic hip arthritis.

Exclusion Criteria:

* DDH

Ages: 1 Week to 15 Years | Sex: All
Age Groups: Child
Study Population: Neonates, infants and children presented with suspected septic hip arthritis.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
To describe the ultrasound abnormalities seen in Patients with septic hip arthritis. | Baseline
  To evaluate:
  1. Synovial membrane thickness .
  2. Synovial membrane vascularity.
  3. Presence of a joint effusion.
  4. Presence of a joint loculation.
  5. Presence of a joint erosions.

IPD SHARING:
Plan to Share IPD: Undecided